CLINICAL TRIAL: NCT02735499
Title: Bladder Instillation of Botox With EMDA for OAB - a Pilot Study
Brief Title: Instillation of Botox in the Bladder in Women With Overactive Bladder (OAB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital of Vestfold (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Dr Hjalmar A Schiotz, MD, PhD, Senior consultant gynecologist, The Hospital of Vestfold
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Botox instillation study
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Overactive Bladder
Keywords: onabotulinum toxin A; Urinary bladder; EMDA; iontophoresis; electrophoresis; Urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — onabotulinum toxin A; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with Botox (Experimental): Onabotulinum toxin A. 200 units of Botox installed into the bladder by catheter.
  Interventions: Drug: onabotulinum toxin A

INTERVENTIONS:
Drug: onabotulinum toxin A — Onabotulinum toxin A is installed into the bladder and EMDA (Electromotive Drug Application) is applied for 30 minutes
  Other Names: Botox

SUMMARY:
Instillation treatment with onabotulinumtoxin A (BOTOX®) in the urinary bladder

DETAILED DESCRIPTION:
Pilot study to evaluate the effect of instillation treatment with onabotulinumtoxin A (BOTOX®) in the urinary bladder using Electromotive Drug Application (EMDA) in women with overactive bladder.

15 women with therapy-resistant OAB will be included. All patients must be qualified for conventional cystoscopic Botox injection. The study is not randomized or blinded. Follow-up time is six months with voiding charts and three questionnaires (Urinary Distress Inventory-6 (UDI-6), Incontinence Impact Questionnaire-7 (IIQ-7), International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI SF) as well as a satisfaction with treatment Visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed
* OAB/urgency incontinence of at least 3 months duration
* Conservative treatment (medicines, electrical stimulation) has been tried without sufficient benefit
* There is indication for cystoscopic injection treatment with Botox®
* More than 3 months since any previous treatment with Botox®
* Detrusor overactivity documented by cystometry is desirable, but not obligatory

Exclusion Criteria:

* Age below 18 years
* Mixed incontinence with predominant stress component
* Insufficient understanding of Norwegian and / or unable to fill out the necessary forms
* Ongoing urinary tract infection (UTI) (defined as positive urine stix (nitrite and leucocytes) with symptoms of UTI) must be treated before inclusion.
* Any contraindication stated in the Summary of product characteristics (SPC) for Botox

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in number of leakage episodes | 24 hours
  Measured with a 24-hour voiding chart

SECONDARY OUTCOMES:
Change in grams leakage | 24 hours
  Measured with a 24-hour voiding chart
Change in number of voids | 24 hours
  Measured with a 24-hour voiding chart
Change in mean voided volume | 24 hours
  Measured with a 24-hour voiding chart
Change in Urinary Distress Inventory-6 score (UDI-6) | 6 months
  Questionnaire
Change in Incontinence Impact Questionnaire-7 score (IIQ-7) | 6 months
  Questionnaire
Change in International Consultation on Incontinence Questionnaire-Short Form score (ICIQ-SF) | 6 months
  Questionnaire
Change in flow rate | 4 weeks
  Measured by flowmetry

CONTACTS AND LOCATIONS:
Overall Officials: Hjalmar A Schiotz, MD, PhD, Principal Investigator — Vestfold Hospital
Locations (1):
- Dept of Ob/Gyn, The Hospital of Vestfold, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duthie JB, Vincent M, Herbison GP, Wilson DI, Wilson D. Botulinum toxin injections for adults with overactive bladder syndrome. Cochrane Database Syst Rev. 2011 Dec 7;2011(12):CD005493. doi: 10.1002/14651858.CD005493.pub3. PMID 22161392
- [Background] Kajbafzadeh AM, Ahmadi H, Montaser-Kouhsari L, Sharifi-Rad L, Nejat F, Bazargan-Hejazi S. Intravesical electromotive botulinum toxin type A administration--part II: Clinical application. Urology. 2011 Feb;77(2):439-45. doi: 10.1016/j.urology.2010.06.003. Epub 2010 Aug 30. PMID 20800886
- [Result] Schiøtz HA, Mai HT, Zabielska R. Intravesical Electromotive Botulinum Toxin in Women with Overactive Bladder - a pilot study. AJGO 2017; 2: 4-10. https://www.arcjournals.org/pdfs/ajgo/v2-i2/2.pdf
- See also: Final article — http://dx.doi.org/10.20431/2456-0561.0202002